CLINICAL TRIAL: NCT04290286
Title: Interdisciplinary, Internet-based Trans Health Care (i2TransHealth): A Randomized Controlled Trial
Brief Title: i2TransHealth: Interdisciplinary, Internet-based Trans Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Timo Nieder, PI: Timo Nieder, PhD ECPS, Head of Outpatient Unit for Sexual Health and Transgender Care, Institute for Sex Research, Sexual Medicine and Forensic Psychiatry (Co-PI: Arne Dekker, PhD, Peer Briken, MD FECSM Prof)), Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: i2TransHealth
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Gender Dysphoria; Gender Identity Disorder; Transsexualism; Gender Identity; Gender Incongruence
MeSH Terms: conditions — Gender Dysphoria; Transsexualism

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): TGD people (n = 82) receive 4 months of e-health intervention according to the i2TransHealth model of care (intervention group)
  Interventions: Other: i2TransHealth
- waiting group (No Intervention): TGD people (n = 82) wait 4 months until they are offered regular care (waiting group), which can include video consultation

INTERVENTIONS:
Other: i2TransHealth — i2TransHealth: online intervention for TGD people
  Arms: intervention group

SUMMARY:
i2TransHealth is a randomized controlled trial that investigates the outcomes of an internet-based health care approach for transgender and gender diverse (TGD) people. As a health services research project, i2TransHealth aims at reducing the structural disadvantage for TGD people [people with transsexualism (TS: ICD-10), gender incongruence (GIC: ICD-11) and/or gender dysphoria (GD: DSM-5)] living in areas lacking specialized transition-related treatment.

Located at the Institute for Sex Research and in cooperation with the Interdisciplinary Transgender Health Care Center Hamburg (ITHCCH), both University Medical Center Hamburg-Eppendorf (UKE), i2TransHealth is an innovative intervention including video consultation and a 1:1 chat with clinical psychologists. By cooperating with the ITHCCH, general physicians and psychiatrists provide first and local access to the specialized treatment provided by the UKE.

In the intervention group, the study participants are invited to use the i2TransHealth e-health platform including a video consultation hour every two weeks and a messenger between the video-meetings. In addition, they have the opportunity to receive medical support close to their home by licensed GPs and psychiatrists according to their needs (especially in case of a somatic or mental health crisis). The waiting group participants will be able to go forward with transition-related care after four months of study participation, as part of regular care.

The primary outcome measure is a reduced symptomatology for TGD people (BSCL). Secondary outcome parameters include quality of life and patient satisfaction as well as healthcare-related costs and cost-effectiveness. Finally, based on a longitudinal design, it will be assessed if the physicians improve their TGD-related expertise by cooperating within the i2TransHealth-network.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Gender different from their assigned sex at birth
* resident at least 50 km outside Hamburg
* present themselves with treatment needs (TS/GD) to one of the participating physicians in the i2TransHealth network, or direct contact with institute and/or e-health platform
* receive the suspected diagnosis TS/GD during an initial interview in the UKE
* can operate the video chat cognitively, verbally and auditory
* Able to read, speak, and understand German
* Written informed consent after written and oral information

Exclusion Criteria:

* Under 18 years of age
* Missing informed consent
* Unable to speak German
* Indication for inpatient treatment, e.g. due to acute psychotic symptoms (self-report, Prodromal Questionnaire, PQ-B) or severe depressive symptoms (self-report, BDI-II ≥ 29)
* Acute suicidal tendencies
* Decrease in intelligence (IQ below 70)
* Acute drug intoxication
* Failure to meet technical requirements (no Internet access, lack of IT knowledge)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Symptom burden according to BSI-18 | Change from Baseline Mental Health Symptoms to the point of time after online intervention (Baseline + 4 months)
  References:
  Franke, G. H. (2000). Franke, G.H. (2000). BSI. Brief Symptom Inventory - Deutsche Version. Manual. Göttingen: Beltz.

SECONDARY OUTCOMES:
Quality of Life (physical health, psychological health, social relationships, and environment) | Change from Baseline QoL to the point of time after online intervention (Baseline + 4 months)]
  QoL is measured using the WHOQOL-BREF (WHO, 1998).
  References:
  Angermeyer, M. C., Kilian, R., & Matschinger, H. (2000). WHOQOL - WHOQOL-100 und WHOQOL-BREF. Handbuch für die deutschsprachigen Versionen der WHO Instrumente zur Erfassung von Lebensqualität.
  WHO (1998). Development of the World Health Organization WHOQOL-BREF quality of life assessment. Psychological medicine, 28(3), 551-558.
Treatment satisfaction according to modified version ZUF-8 | Treatment satisfaction at the point of time after online intervention (4 months after admission to studies)
  References:
  Schmidt, J., Lamprecht, F., & Wittmann, W. W. (1989). Zufriedenheit mit der stationären Versorgung. Entwicklung eines Fragebogens und erste Validitätsuntersuchungen. [Satisfaction with inpatient care: Development of a questionnaire and first validity assessments.]. PPmP: Psychotherapie Psychosomatik Medizinische Psychologie, 39(7), 248-255.
Direct or indirect costs and productivity losses by persons with TS/GD in comparison to the German general population (via CSSRI) | Change from Baseline to the point of time after online intervention (Baseline + 4 months)
  References:
  Chisholm, D., Knapp, M. R. J., Knudsen, H. C., Amaddeo, F., Gaite, L., Wijngaarden, B. van, & Group, E. S. (2000). Client Socio-Demographic and Service Receipt Inventory - European Version: Development of an instrument for international research: EPSILON Study 5. The British Journal of Psychiatry, 177(S39), s28-s33. https://doi.org/10.1192/bjp.177.39.s28
Health-related quality of life (via EQ-5D-5L): quality-adjusted life years (QALYs) | Change from Baseline to the point of time after online intervention (Baseline + 4 months)
  References:
  Herdman, M., Gudex, C., Lloyd, A., Janssen, MF., Kind, P., Parkin, D., … Badia, X. (2011). Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Quality of Life Research, 20(10), 1727-1736. https://doi.org/10.1007/s11136-011-9903-x
Knowledge increase of the cooperating physicians on trans health care (via VSE) | Change from Baseline to the point of time after study completion (Baseline + 18 months)
  References:
  Raupach, T., Schiekirka, S., Münscher, C., Beißbarth, T., Himmel, W., Burckhardt, G., & Pukrop, T. (2012). Implementierung und Erprobung eines Lernziel-basierten Evaluationssystems im Studium der Humanmedizin. GMS Zeitschrift für medizinische Ausbildung, 29(3), 1-14.
Satisfaction of the cooperating physicians with the support in the i2TransHealth network (via modified version ZUF-8) | Satisfaction at the point of time after study completion (18 months)
  References:
  Schmidt, J., Lamprecht, F., & Wittmann, W. W. (1989). Zufriedenheit mit der stationären Versorgung. Entwicklung eines Fragebogens und erste Validitätsuntersuchungen. [Satisfaction with inpatient care: Development of a questionnaire and first validity assessments.]. PPmP: Psychotherapie Psychosomatik Medizinische Psychologie, 39(7), 248-255.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmidt F, Renner J, Schroder SI, Pregartbauer L, Dekker A, Nieder TO. Enabling and hindering aspects of the i(2)TransHealth e-health intervention for transgender and gender diverse people in Germany: a qualitative process evaluation. BMC Health Serv Res. 2026 Jan 24. doi: 10.1186/s12913-026-14026-y. Online ahead of print. PMID 41580775
- [Derived] Grochtdreis T, Konnopka A, Renner J, Konig HH, Dekker A, Briken P, Nieder T, Dams J. Excess costs of transgender and gender-diverse people with gender incongruence and gender dysphoria compared with people from the general population in Germany: a secondary analysis using data from a randomised controlled trial and a representative telephone survey. BMJ Open. 2025 Apr 9;15(4):e089663. doi: 10.1136/bmjopen-2024-089663. PMID 40204312
- [Derived] Nieder TO, Renner J, Sehner S, Pepic A, Zapf A, Lambert M, Briken P, Dekker A. Effect of the i2TransHealth e-health intervention on psychological distress among transgender and gender diverse adults from remote areas in Germany: a randomised controlled trial. Lancet Digit Health. 2024 Dec;6(12):e883-e893. doi: 10.1016/S2589-7500(24)00192-4. Epub 2024 Oct 16. PMID 39419729
- [Derived] Nieder TO, Renner J, Zapf A, Sehner S, Hot A, Konig HH, Dams J, Grochtdreis T, Briken P, Dekker A. Interdisciplinary, internet-based trans health care (i(2)TransHealth): study protocol for a randomised controlled trial. BMJ Open. 2022 Feb 1;12(2):e045980. doi: 10.1136/bmjopen-2020-045980. PMID 35105559
- See also: https://www.i2transhealth.de/english-landing-page/ — https://www.i2transhealth.de/